## **RESEARCH PROPOSAL**

**Title**: Immediate Effect Of Standing Trunk Extension Postures On Spinal Height And Clinical Outcome Measures In Low Back Pain: A Randomized Clinical Trial

# Investigators:

Jean-Michel Brismée, PT, ScD - PI Jeremy Harrison, PT, DPT Phillip S. Sizer, PT, PhD

Clinical Musculoskeletal Research Laboratory, Center for Rehabilitation Research, School of Health Professions, TTUHSC, Lubbock, TX, USA

# TABLE OF CONTENTS

| ABSTRACT | 4 |
|---------------------------|----|
| LIST OF FIGURES | 5 |
| LIST OF ABBREVIATIONS | 6 |
| BACKGROUND | 7 |
| PURPOSE, AIMS, VALUES | 12 |
| RESEARCH QUESTIONS | 13 |
| HYPOTHESES | 13 |
| COMPARISON VARIABLES | 14 |
| Independent Variables | 14 |
| Dependent Variables | 15 |
| Relationship Variables | 15 |
| METHODS | 16 |
| Research Design | 16 |
| Pre-Study Approvals | 16 |
| Subjects | 16 |
| Testing Sequence | 17 |
| DATA ANALYSIS | 22 |
| RESEARCH PROJECT TIMELINE | 25 |
| REFERENCES | 26 |
| APPENDICES | 41 |

### **ABSTRACT**

**Background:** Standing trunk extension postures have been used for many years as a mechanical approach to low back pain (LBP), sometimes directed by therapeutic intervention, sometimes subconsciously performed by patients to relieve LBP. However, no study to date has investigated the effect of standing trunk extension postures on spinal height and clinical outcome measures.

**Objective:** The purpose of this study will be to evaluate in subjects with LBP following a period of trunk loading, how spinal height and/or pain, symptoms' centralization, and function outcome measures respond to: (1) standing repetitive trunk extension posture; and (2) standing sustained trunk extension posture. Lumbar range of motion (ROM) achieved during these two trunk extension postures will be compared to spinal height and outcome measures.

**Methods:** A pre-test, post-test comparison group design (randomized clinical trial) will be used to determine how spinal height changes in response to sustained and repetitive standing trunk extension after a period of spinal loading. The study will use a 2 (between subjects – type of trunk extension: sustained vs. repetitive) x 3 (within subjects - time: before vs. after vs. 2 weeks after intervention) mixed design to evaluate the effects of sustained and repetitive trunk extension in standing on spinal height, pain, symptoms' centralization and function.

**Statistical Analysis:** A 2(Strategy) X 3(Time) mixed ANOVA will be used to statistically identify significant interactions and main effects for spinal height, pain and function outcome measures. Post-hoc pairwise comparisons will be used to locate significant differences between the different conditions (Time). Significance will be set at  $\alpha$  = 0.05. Pearson product-moment correlations will be used to measure correlations between lumbar ROM in relation to spinal height and outcome measures. The Kruskal-Wallis 1-factor ANOVA for difference scores will used to determine changes of intensity and location of symptoms following sustained versus repetitive standing trunk extension. Spearman Rank correlation will be used to evaluate the relationship between spinal height changes and changes of pain and location of symptoms for each group.

Word Count: 326

**Key Words**: Standing postures; trunk extension; spinal height change; stadiometer

## **Lay Summary**

Standing back extension postures have been used for many years to treat people with low back pain.

No study to date has investigated the effect of standing back extension postures on trunk height, pain and function.

The **purpose** of this study will be to evaluate in subjects with low back pain how trunk height, pain and function respond to standing repetitive versus sustained trunk extension postures.

**Methods**: A randomized clinical trial will be used to determine how trunk height, low back pain and function change in response to sustained and repetitive standing trunk extension after a period of spinal loading.

**Statistical Analysis** will be used to measure the outcomes.

# LIST OF FIGURES

| Figure 1: Flowchart depicting testing sequence | 31 |
|---|---|
| Figure 2: Starting position for standing trunk extension (repetitive and sustained | 34 |
| Figure 3: Sustained trunk extension position and end position of repetitive trunk extension | |
| Figure 4: Position of subject for spinal height measure in stadiometer unit | 36 |
| Figure 5: Position of subject during spinal loading time in sitting | 37 |
| Figure 6: Home exercise program for repetitive trunk extension group | 38 |
| Figure 7: Home exercise program for sustained trunk extension group | 39 |
| Figure 8: Home instructions for each subject | 40 |

# LIST OF ABBREVIATIONS

| Analysis of Variance | ANOVA |
|-------------------------------------|-------|
| Fear Avoidance Belief Questionnaire | FABQ |
| Intervertebral Disc | IVD |
| Institutional Review Board | IRB |
| Low Back Pain | LBP |
| Numerical Pain Rating Scale | NPRS |
| Range of Motion | ROM |
| Standard Deviation | SD |
| Research Question | RQ |
| Research Hypotheses | RH |
| Independent Variable | IV |
| Dependent Variable | DV |
| Relationship Variable | RV |

### **BACKGROUND**

According to the United States Department of Labor, there were more than one million injuries and illnesses requiring days away from work amongst private industry, state and local government employees. Among these injuries and illnesses, 16.6 % were low back related equating to 191,479 low back injuries requiring days away from work (US Department of Labor, Bureau of Labor Statistics, 2016). An analysis funded by the National Institute of Health found that the cost of pain outweighed the cost of cancer and diabetes by thirty percent. The authors further reported that the annual cost of pharmaceuticals for pain management was \$16.4 billion, and the cost of lumbar surgeries was \$2.9 billion. Pain indirect costs estimates were \$18.9 billion for disability compensation and \$6.9 billion for productivity loss (Gaskin 2011, The Economic Costs of Pain in the United States).

A joint clinical practice guideline developed by the American College of Physicians and the American Pain Society classified low back pain (LBP) into three categories: (1) nonspecific LBP; (2) LBP potentially associated with radiculopathy or spinal stenosis; and (3) LBP potentially associated with another specific spinal cause. Of those three, lumbar intervertebral disc (IVD) herniation is one of the most common spinal degenerative disorders leading to LBP associated with radiculopathy (Chou 2007, Goupille 1998, McCall 2000). In order to better understand the IVD's role in the development or persistence of LBP and spinal stenosis, there have been many stadiometric studies primarily focused on lumbar spinal height changes associated with various positions and movements

(Kourtis 2004; Magnusson 1996; Lazzarini 2014; Simmerman 2011). These studies stem from IVD height preservation in the aging spine. Natural IVD height preservation is so important that the biomedical field has examined the use of growth factors for IVD biologic regeneration (Masuda 2004) in order to more naturally preserve IVD biomechanical and physiological function as opposed to surgical disruption. To further understand IVD functional properties, researchers have studied the IVD hydraulic permeability and the influence that age and/or degeneration have on fluid movement (Gu 1999). The authors reported that with IVD degeneration, the radial permeability of the anulus fibrosus decreased, mainly because of reduced water content. However, the axial and circumferential permeability coefficients increased, mainly due to structural change, leading to greater IVD isotropic permeability behavior (Gu 1999).

Sixty one percent of time in the work and home environment is spent in the standing posture (US Department of Labor, Bureau of Labor Statistics, 2016). Although prolonged weight bearing postures, such as standing and walking, have been associated with decreased spine height (Tyrrell 1985, Puntumetakul et al 2009), some studies reported that seated weight bearing postures could result in spine height gain (Magnusson 1996a). Sustained and repetitive lumbar extension postures frequently occur after periods of prolonged unloading such as sleep. These postures are periodically repeated throughout the day during activities such as standing and walking (US Department of Labor Bureau of Labor Statistics 2016).

People presenting with directional preferences that include lumbar

extension tend to respond well to exercises geared toward trunk extension (Stankovic 1990, Swinkels 2009, Oliveira 2012). Significant and rapid changes in central and distal pain intensity and location have resulted from standing endrange trunk extension in patients with low back and referred pain (Donelson 1991). Additional studies reported that standing back extension exercises resulted in back pain episodes' prevention and decreased back pain in care workers (Matsudaira 2015; Dunsford 2011). Standing exercises have the advantage to be functional and easily performed in work and home settings (Tonosu 2016).

A positive relationship has been found between lumbar extension range of motion (ROM) and the centralization process in patients with LBP (Bybee et al 2009). The centralization phenomenon is part of the clinical examination findings used to identify specific treatment-based classification subgroups. Centralization is characterized by spinal pain and referred symptoms that are progressively abolished in a distal to proximal direction in response to therapeutic interventions including unloading or specific movement strategies (Brennan et al 2006, Laslett et al 2005). The operational definition and measurement techniques for centralization have been laid out in several studies (Aina et al 2004, Werneke et al 2008). A decreased spinal ROM is commonly associated with low back complications, and functional ROM needs to be restored to allow for the return to previous activity levels (Battie 1987, Vaisy 2015). Several methods have been used to increase spinal ROM including static, repeated, passive postures, and proprioceptive neuromuscular facilitation. Both standing and prone lumbar

extension postures are effective for treating low back Dysfunction Syndrome (McKenzie 2003). However, which method is best suited for increasing spinal ROM remains debated (Sady 1982; Nordez 2017). One author found static prone postures to increase ROM more effectively with 30-60 second sustained postures as compared to 15-second postures, but no difference between the effectiveness of 30-second and 60-second postures (Bandy 1994; Page 2012).

Repetitive postures are another method used to increase ROM by elongating shortened connective tissue. The McKenzie classification of Dysfunction Syndrome is defined as the condition in which adaptive shortening of soft tissues and resultant loss of mobility cause pain by stretching shortened tissues that block full end-range movement (Hefford 2008). Poor postural habits, previous trauma and inflammatory or degenerative processes can lead to this dysfunction. These patients can develop contraction, scarring, adherence and adaptive shortening or imperfect repair and pain is felt when the abnormal tissue is stretched.

Treatment of the Dysfunction Syndrome consists of postural correction, along with repeated end-range movements to remodel contracted structures. This intermittent stress is reported to provide an adequate stretching effect and is most effective in the treatment of extension dysfunction (McKenzie 2003). One study found that patients with LBP chose to perform their extension posture for home exercise in standing 80.8 % of the time and only 19.2 % of the time in the prone position, resulting in similar clinical outcomes where both groups showed equal improvements in lumbar extension ROM (Bybee et al 2008).

Previous studies investigated the effects of postures and movements in lying (unloaded) or seated positions on spinal height (Owens 2009, Gerke et al 2010; Pape 2018). These studies primarily focused on spinal height following static patient positioning and showed that both the lying and supported seated positions resulted in mean spinal height gains of 2 to 5 mm. However, most rehabilitation programs focused on LBP prevention and management use both repetitive and/or sustained spinal extension exercises to improve patients' outcomes (Peterson 2015, Surkitt 2012). Such exercises can be performed in lying or standing position. Although patients with acute and recurrent low back and referred pain tend to respond well to directionally preferenced postures (Machado 2006), subjects with chronic symptoms tend to display greater signs of sensitization, biopsychosocial issues (Huysmans 2017), and tend to respond less favorably to directional preferences postures and exercises (Garcia 2017). In order to assess the biopsychosocial effect on clinical outcomes during this study, every subject will complete the Fear Avoidance Belief Questionnaire (FABQ) (Cleland et al 2008).

No study to date has investigated the effects of standing extension postures on spinal height, pain, centralization and function. Therefore, the purposes of this study will be to evaluate in a sample of LBP patients the effect of standing trunk extension, both sustained and repetitive, following a period of spinal loading, on (1) spinal height; (2) pain; (3) symptoms centralization and (4) functional measures.

## PURPOSE, AIMS, VALUES

### Purpose(s):

The purpose of this study is to assess the effect of commonly used standing trunk extension postures on spinal height as well as pain, symptoms' centralization, and function in patients with LBP.

## Aim(s):

Our aim is to better understand the effect of standing sustained and repetitive trunk extensions on spinal height and LBP patients' symptoms intensity, centralization and function. With many patients commonly falling into a directional preference group and responding positively to mechanical spinal input, it is our aim to investigate if such trunk extension postures performed in standing affect spinal height in regard to growth or shrinkage and if these changes are associated with symptoms intensity, centralization and functional alterations.

## Value(s):

No previous study has examined changes in spinal height following standing trunk extension postures and little is known on the effect of such standing postures on spinal height. The results of this study could impact rehabilitation programs that include standing trunk extension as a means of therapeutic intervention. This is valuable especially in aging population with degenerated IVD's, loss of IVD height and propensities toward spinal stenosis, as we do not know if those subjects with directional preferences toward spinal extension could use standing trunk extension postures at home or in the work

environment to grow and/or prevent spinal shrinkage.

RESEARCH QUESTIONS, HYPOTHESES AND VARIABLES

**Research Question(s)** (RQs)-This project aims to answer the following research questions:

- 1. RQ 1: Does sustained and repetitive standing trunk extension following a period of spinal loading effect spinal height, pain, centralization and function testing outcomes immediately and two weeks following the interventions in patients with LBP?
- 2. RQ 2: Following a period a spinal loading, is there a difference in spinal height, pain, centralization and function testing outcome *changes* immediately and two weeks following sustained and repetitive standing trunk extension postures in patients with LBP?
- 3. RQ 3: Is there a correlation between the degree of trunk extension during standing lumbar extension posture and spinal height, pain, centralization and function testing outcomes *changes* immediately and two weeks following the interventions in patients with LBP?

**Research Hypotheses- (RH)**This student has devised the following research hypotheses:

 RH 1: It is expected that following a period of trunk loading, both sustained and repetitive trunk extension postures in standing will result in increased spinal height, reduced pain, enhanced centralization and

Harrison, Research Proposal

function testing outcomes immediately and two weeks following the

interventions in patients with LBP.

2. RH 2: It is expected that following a period of trunk loading, sustained

standing trunk extension posture in standing will result in greater spinal

height gain as compared to repetitive standing trunk extension postures,

while repetitive standing trunk extension postures will result in greater

improvements in pain, centralization and function testing outcomes as

compared to sustained standing trunk extension postures immediately

and two weeks following the interventions.

3. RH 3: It is expected that following a period of trunk loading, there will be a

positive correlation between the degree of trunk extension during

standing trunk extension posture and spinal height, centralization, pain

and function testing outcomes changes immediately and two weeks

following the interventions in patients with LBP.

Comparison Variables

Independent Variable(s)-The student plans to use the following Independent

variable(s) (IV)

1. IV1: Trunk extension

a. IV1: sustained

b. IV2: repetitive

2. IV2: Time

14

- a. IV1: before
- b. IV2: after (immediately)
- c. IV3: after 2 weeks

**Dependent Variable(s)**-The Student plans to measure the following dependent variable(s) (DV)

- 1. DV1: Spinal height using stadiometer (ratio scale).
- DV2: Pain rating using numerical pain rating scale (NPRS) (ordinal scale).
- 3. DV3: Centralization (ordinal) using body diagram.
- 4. DV4: Modified Oswestry Pain Disability Questionnaire (ordinal scale)

## **Relationship Variable(s)-** (RV) (if applicable)

- 1. RV1: Degree of spinal extension (ratio)
- 2. RV2: Spinal height using stadiometer (ratio scale).
- RV3: Pain rating using numerical pain rating scale (NPRS) (ordinal scale).
- 4. RV4: centralization (ordinal).
- 5. RV5: Modified Oswestry Pain Disability Questionnaire (ordinal scale)

### **METHODS**

## Research Design(s)

A pre-test, post-test comparison group design (randomized clinical trial) will be used to determine how spinal height changes in response to sustained and repetitive standing trunk extension after a period of spinal loading. The study will use a 2 (between subjects – type of trunk extension: sustained vs. repetitive) x 3 (within subjects - time: before vs. after vs. 2 weeks after) mixed design to evaluate the effects of sustained and repetitive trunk extension in standing on spinal height, pain, centralization and function outcome measures.

# **Pre-study Approvals**

The study will be submitted to the Texas Tech University Health Sciences

Center Institutional Review Board (IRB) for approval. The trial will then be
registered at https://clinicaltrials.gov.

### Subjects / Specimens

Systematic consecutive sampling of up to 100 subjects with LBP (40 subjects completing both days of data collection) attending "Sports medicine and Physical therapy clinic" in Fredericksburg (Texas) as patients or for the purpose of health and wellness will be recruited. Flyers will also be posted at physician offices and the general Fredericksburg community and surrounding areas to inform subjects about the study (Appendix A).

Inclusion Criteria: (1) Ability and willingness to come twice to the clinic for approximately 60 minutes each; (2) Subjects with LBP and directional preference

in back extension; (3) Age 18-80 (Yarznbowicz et al 2018); (4) Ability to stand for 5 minutes; (5) Ability to sit for 10 minutes; and (6) Low back pain on Numerical Pain Rating scale (NPRS) of at least 2/10 and less or equal to 9/10 (Ferreira-Valente 2011).

Exclusion Criteria: (1) Pregnancy by subject report; (2) history of back surgery or spinal fractures within the last six months; (3) history of spinal fusion or physician's diagnosis of spinal instability; (4) current history of acute systemic infection, active inflammatory disease, or malignancy; (5) subjects engaged in legal/compensation claims for their back symptoms; and (6) subjects unable to understand or speak English.

## **Testing Sequence**

Subjects will be asked to attend two physical therapy sessions over approximately a 60-minute period each to complete the study.

## Session 1

Participants will complete a pre-screening questionnaire regarding inclusion (Appendix B). Each subject will watch an audio-visual power point presentation explaining the study, test procedures and describing the interventions (standing repetitive trunk extension and standing sustained trunk extension). Written informed consent will be obtained. To determine directional preference, the investigator (JH) will use the guidelines set forth in the directional preference definition (Werneke 2011) and based off of standards set forth in randomized clinical trials (May et al 2008). Directional preference has been

defined as either (1) a specific direction of trunk movement or posture noted during the physical examination or (2) a specific easing factor reported by the patient during the subjective history that alleviates or decreases the patient's pain, with or without the pain having changed location and/or increased the patient's lumbar range of motion (Werneke 2011). A questionnaire including pertinent medical history will be completed (Appendix C). Subjects will complete (1) a Numerical Pain Rating Scale (NPRS) to rate their current, minimum, maximum and average LBP over the last two days (Ferreira-Valente MA 2011) as well as paresthesia signs/symptoms intensity (Appendix D); (2) Body Diagram for indicating location of symptoms (Appendix E); (3) Modified Oswestry low back pain questionnaire (Fritz 2001) (Appendix F); (4) Fear Avoidance Belief Questionnaire (Cleland et al 2008) (Appendix G). A researcher will record subject's height and weight. A Flow chart illustrates study sequence in details (Figure 1).

If the subject meets criteria for inclusion in the study, the subject will complete a familiarization procedure to determine the consistency to reposition themselves in the stadiometer. Subjects able to reposition themselves in the stadiometer with a SD of 1.3mm or less for five consecutive measurements (Stothart et al 2000; Gerke et al 2011; Owens et al 2009) will be included in the study. The digital display will be covered to blind the researcher performing the measurements. The data will be automatically recorded by the stadiometer and manually downloaded to a laptop computer.

At the beginning of data collection, a randomization plan generator

(http://www.randomization.com ) will assign each subject to one of two interventions: (1) standing repetitive trunk extension at a rate of 10 per 45 seconds (Figure 2), repeated five times with 15-second rest breaks; or (2) standing sustained trunk extension for 5 x 45 seconds with 15-second rest breaks (Figure 3). Each subject will complete one intervention. The intervention number assigned will be recorded by the subject next to their name to allow blinding of the investigator as to which intervention the subject is assigned to. The subject will undergo the test sequence after a 10-minute period of trunk unloading in a supine posture to ensure spinal height is normalized, head in neutral posture, knees supported over a small bolster pillow, hands placed on the abdomen (Kourtis et al 2004; Magnusson et al 1996a; Gerke et al 2011; Owens et al 2009). The subject will reposition on the stadiometer and spinal height will be measured after a relaxed exhalation (Measurement 1) (Figure 4). The subject then will undergo a five-minute period of loaded upright sitting with a 4.5kg bag secured on each shoulder and spinal height will be measured (Measurement 2) (Figure 5) (Kourtis et al 2004; Owens et al 2009; Gerke et al 2011). As continued spinal height reduction has been demonstrated following loaded sitting, the subject will undergo an additional five minutes sitting without load and spinal height will be measured (Measurement 3) (Kourtis et al 2004; Owens et al 2009; Gerke et al 2011). Inclinometers will be used to take an initial measure of each subject trunk extension prior to intervention. The subject will then undergo one intervention for 5 minutes as previously described, according to the randomization assignment. In order to determine how sustained and repetitive

interventions related in terms of change in spinal height, the time to perform the sustained lumbar posture matches the time necessary to perform the repetitive lumbar extension postures.

The subject will reposition on the stadiometer and spinal height will be measured (Measurement 4). Trunk extension will be measured to determine the strength of correlations between the degree of trunk extension during standing trunk extension posture and spinal height, pain and centralization testing outcomes changes (MacDermid et al 2015). The subject will score their low back and lower extremity symptoms using NPRS (Ferreira-Valente MA 2011), and map their pain on a body pain diagram (Appendix E) prior to intervention, immediately after and 2-week following the intervention to determine pain rating and centralization of symptoms (Simmerman et al 2011). The principal investigator will apply a numeric overlay template to the patient's body diagrams to document the most distal pain location scores between 1 and 6 (Appendix I). Higher score will indicate a more distal symptoms' location.

## Home instructions

Subjects will be instructed to continue to use their medications, including medications aimed at decreasing their pain, as prescribed by their primary healthcare provider and not to change them during the follow-up two-week period. A sheet including home exercise instructions will be provided to each patient. Instructions will include repetitive or sustained trunk extension based on random group assignment, performed approximately 5 times per day. Each subject will complete a sheet recording home exercise compliance upon arrival in

session 2 (Appendix I).

## Session 2

Subjects will complete: (1) a NPRS to rate their current, minimum, maximum and average LBP over the last two days as well as paresthesia signs/symptoms intensity (Appendix D); (2) Body Diagram for indicating location of symptoms (Appendix E) (3) Modified Oswestry low back pain questionnaire (Fritz 2001) (Appendix F); (4) Fear Avoidance Belief Questionnaire (Cleland et al. 2008) (Appendix G). Each subject will then complete a familiarization procedure to determine the consistency to reposition themselves in the stadiometer as described in session 1. The subject will undergo a 10-minute period of trunk unloading in a supine posture to ensure spinal height is normalized as described in session 1. The subject will reposition on the stadiometer and spinal height will be measured after a relaxed exhalation (Measurement 1) (Figure 4). The subject then will undergo a five-minute period of loaded upright sitting with a 4.5kg bag secured on each shoulder and spinal height will be measured (Measurement 2) (Figure 5). The subject will then undergo an additional five minutes sitting without load and spinal height will be measured (Measurement 3). Inclinometers will be used to take an initial measure of each subject trunk extension prior to intervention. The subject will then undergo the same intervention as in session 1 for 5 minutes as previously described (standing repetitive trunk extension or standing sustained trunk extension). The subject will reposition on the stadiometer and spinal height will be measured (Measurement 4). Trunk extension will be measured to determine the strength of correlations between the degree of trunk extension during standing trunk extension posture and spinal height, pain and centralization testing outcomes changes (MacDermid et al 2015). The subjects will then score their low back and lower extremity symptoms using NPRS (Ferreira-Valente MA 2011), and *map their pain* on a body pain diagram (Appendix H).

## **Investigator Blinding**

One investigator will be involved with data collection. The investigator,
Jeremy Harrison, PT, DPT will carry out inclinometer measurements of lumbar
and sacral posture, supervised positioning in the stadiometer and stadiometric
measurements. The investigator will be blinded to the intervention (each subject
will receive a hidden random number and will perform independently the
intervention in a treatment room) and the stadiometric measurements during the
experiment. He will also be responsible for assigning subjects to their initial
groups, supervising the subjects' positioning in the different standing postures
and confirming that a stadiometer reading is recorded on an Excel spreadsheet.

## **Subjects Compensation**

Subjects will receive a one-month free membership to Hill Country

Memorial Wellness Center in Fredericksburg, Texas if they consent to participate in the study.

## Subjects Charges

There will be no charge for the two physical therapy sessions, including

examination and intervention. Following the two intervention sessions, subjects referred by primary care providers (physicians, chiropractors, nurse practitioners, physician assistants) to physical therapy for LBP will have the choice to receive standard care and be charged for physical therapy intervention.

## Confidentiality and data protection

Electronic Transmission of Personally Identifiable Information (PII) and Protected Health Information (PHI) will be followed and computer device has been encrypted (password protected). Excel spreadsheet will be used to store the data. No Personally Identifiable Information will be retained in the Excel spreadsheet where the data will be stored.

## **Data Analysis**

Descriptive and inferential statistics will be used utilizing SPSS 23.0 for Windows (SPSS, Chicago, IL).

- 1. Descriptive analyses: Descriptive statistics including mean, median, mode, standard deviation, minimum and maximum values, frequency counts will be collected for age, height, weight, body mass index, pain, centralization, function (Oswestry Low Back Pain Disability Questionnaire), Fear Avoidance Beliefs Questionnaire, spinal height, and spinal height changes after repetitive and sustained standing trunk extension after a period of spinal loading.
- 2. **Inferential analyses:** Levene's test and Shapiro-Wilk test of normality will used to test for variance and distribution of measurements of spinal height,

changes in spinal height, degrees of spinal extension, pain, and function outcomes.

For experimental hypothesis 1, a paired-t-test (or Wilcoxon sign-rank test if the data do not meet assumptions for parametric inferential statistics) will be used to assess differences in spinal height, centralization and pain outcomes improvements following sustained and repetitive trunk extension postures.

For experimental hypothesis 2, 2 (between subjects - type of trunk extension: sustained vs. repetitive) x 3 (within subjects - time: before, immediately after and 2-week after) mixed ANOVA's will examine differences in (1) spinal height; (2) pain; and (3) function outcomes, as a result of sustained and repetitive standing trunk extension after a period of spinal loading. Post hoc paired t-tests will explore further for significant differences in spinal height, pain and function outcomes between the six conditions.

Experimental hypothesis 3 will be tested with Pearson product-moment correlations to determine the strength of correlations between the degree of trunk extension during standing trunk extension posture and spinal height, pain and function, outcomes changes in patients with LBP.

Spearman's Rank Order correlation will be used to determine the strength of the correlation between centralization and the degree of trunk extension posture in standing.

Alpha level will be set at 0.05 for significance for all tests and Bonferroni corrections performed as needed.

### **REFERENCES**

- 1. Aina A, May S, Clare H. The centralization phenomenon of spinal symptoms a systematic review. Man Ther. 2004;9:134-143.
- 2. Alexander LA, Hancock E, Agouris I, Smith FW, MacSween A. The response of the nucleus pulposus of the lumbar intervertebral discs to functionally loaded positions. Spine. 2007;32:1508-1512.
- 3. Battie MC, Bigos SJ, Sheehy A, Wortley MD. Spinal flexibility and individual factors that influence it. Phys Ther. 1987;67:653-658.
- 4. Brennan G, Fritz J, Hunter S, Thackeray A, Delitto A, Erhard R. Identifying subgroups of patients with acute/subacute "nonspecific" low back pain: results of randomized clinical trial. Spine. 2006;31:623-631.
- 5. Bybee RF, Mamantov J, Meekins W, Witt J, Byars A, Greenwood M. Comparison of two stretching protocols on lumbar spine extension. J Back Musculoskeletal Rehabil. 2008;21:153-159.
- 6. Bybee RF, Olsen DL, Cantu-Boncser G, Allen HC, Byars A. Centralization of symptoms and lumbar range of motion in patients with low back pain. Physiother Theory Pract. 2009;25:257-267.
- 7. Chou R, Qaseem A, Snow V, Casey D, Cross JT Jr, Shekelle P, Owens DK; Clinical Efficacy Assessment Subcommittee of the American College of Physicians; American College of Physicians; American Pain Society Low Back Pain Guidelines Panel. Diagnosis and treatment of low back pain: a joint clinical practice guideline from the American College of Physicians and the American Pain Society. Ann Intern Med. 2007;147:478-491.
- 8. Cleland JA, Fritz JM, Brennan GP. Predictive validity of initial fear avoidance beliefs in patients with low back pain receiving physical therapy: is the FABQ a useful screening tool for identifying patients at risk for a poor recovery? Eur Spine J. 2008;17:70-79.
- Donelson R, Grant W, Kamps C, Medcalf R. Pain response to sagittal endrange spinal motion. A prospective, randomized multicentered trial. Spine. 1991;16:206-212.
- 10. Dunsford A, Kumar S, Clarke S. Integrating evidence into practice: Use of McKenzie-based treatment for mechanical low back pain. J Multidiscip Healthc. 2011;4:393-402.
- 11. Ferreira-Valente MA, Pais-Ribeiro JL, Jensen MP. Validity of four pain intensity rating scales. Pain. 2011;152:2399-2404.
- 12. Fritz JM, Irrgang JJ. A comparison of a modified Oswestry Low Back Pain Disability Questionnaire and the Quebec Back Pain Disability Scale. Phys Ther. 2001;81:776-788.

- 13. Garcia AN, Costa LDCM, Hancock MJ et al. McKenzie Method of Mechanical Diagnosis and Therapy was slightly more effective than placebo for pain, but not for disability, in patients with chronic non-specific low back pain: a randomized placebo controlled trial with short and longer term follow-up. Br J Sports Med. 2017;52:594-600.
- 14. Gerke DA, Brismee JM, Sizer PS, Dedrick GS, James CR. Change in spine height measurements following sustained mid-range and end-range flexion of the lumbar spine. Appl Ergon. 2011;42:331-336.
- 15. Goupille P, Jayson MI, Valat JP and Freemont AJ. The role of inflammation in disk herniation- associated radiculopathy. Semin Arthritis Rheum. 1998;28:60-71.
- 16. Gu WY, Mao XG, Foster RJ, Weidenbaum M, Mow VC, Rawlins BA. The Anisotropic Hydraulic Permeability of Human Lumbar Anulus Fibrosus. Spine. 1999;24:2449-2455.
- 17. Hefford C. McKenzie classification of mechanical spinal pain: Profile of syndromes and directions of preference. Man Ther. 2008;13:75-81.
- 18. Huysmans E, Ickmans K, Van Dyck D et al. Association Between Symptoms of Central Sensitization and Cognitive Behavioral Factors in People With Chronic Nonspecific Low Back Pain: A Cross-sectional Study. J Manipulative Physiol Ther. 2017;17:30151-3.
- 19. Johannaber K, Fathallah FA. Spinal disc hydration status during simulated stooped posture. Work; 2012;41:2384-6.
- 20. Kourtis D, Magnusson ML, Smith F, Hadjipavlou A, Pope MH. Spine height and disc height changes as the effect of hyperextension using stadiometry and MRI. lowa Orthop J. 2004;24:65-71.
- 21. Laslett M, Oberg B, Aprill C, McDonald B, Centralization as a predictor of provocation discography results in chronic low back pain, and the influence of disability and distress on diagnostic power. Spine J. 2005;5:370-380.
- 22. Lazzarini M, Brismee JM, Owens SC, Dedrick GS, Sizer PS. Spinal height change in response to sustained and repetitive prone lumbar extension after a period of spinal unloading. J Manipulative Physiol Ther. 2014;37(8):586-592.
- 23. Lewis SE, Fowler NE. Changes in intervertebral disc dimensions after a loading task and the relationship with stature change measurements. Arch Phys Med Rehabil. 2009;90:1795-9.
- 24. Machado LA, de Souza Mv, Ferreira PH, Ferreira ML. The McKenzie method for low back pain: a systematic review of the literature with a meta-analysis approach. Spine. 2006;31:254-262.

- 25. MacDermid JC, Arumugam V, Vincent JI, Payne KL, So AK. Reliability of three landmarking methods for dual inclinometry measurements of lumbar flexion and extension. BMC Musculosketal Disor. 2015;16:121.
- 26. Magnusson ML, Aleksiev AR, Spratt KF, Lakes RS, Pope MH. Hyperextension and spine height changes. Spine. 1996;21:2670-5.
- 27. Magnusson M, Hult E, Lindstrom I, Lindell V, Pope M, Hansson T. Measurement of time-dependent height-loss during sitting. Clinical Biomech. 1990;5:137-142.
- 28. Magnusson M, Pope M. Body height changes with hyperextension. Clin Biomech (Bristol, Avon). 1996;11(4):236-238.
- 29. Masuda K, Oegema TR Jr, An HS. Growth factors and treatment of intervertebral disc degeneration. Spine. 2004;29:2757-2769.
- 30. Matsudaira K, Hiroe M, Kikkawa M, Sawada T, Suzuki M, Isomura T, Oka H, Hiroe K, Hiroe K. Can standing back extension exercise improve or prevent low back pain in Japanese care workers? J Man Manip Ther. 2015;23(4):205-9.
- 31. May S, Donelson R. Evidence-informed management of chronic low back pain with the McKenzie method. Spine J. 2008;8:134-141.
- 32. McCaffrey L, LeFebvre R. Directional Preference Protocol: Centralizing Low Back and Leg Pain. WSCC Clinics. 2008:1-12.
- 33. McCall IW. Lumbar herniated disks. Radiol Clin North Am 2000;38:1293-1309.
- 34. McKenzie RA, May S. The Lumbar Spine Mechanical Diagnosis and Therapy, 2<sup>nd</sup> ed. Spinal Publications Ltd. 2003;647-667.
- Nordez A, Gross R, Andrade R et al. Non-Muscular Structures Can Limit the Maximal Joint Range of Motion during Stretching. Sports Med. 2017;47:1925-1929.
- 36. Oliveira VC, Ferreira PH, Maher CG, Pinto RZ, Refshauge KM, Ferreira ML. Effectiveness of self-management of low back pain: Systematic review with meta-analysis. Arthri Care Res. 2012;64:1739-1748.
- 37. Owens SC, Brismee JM, Pennel PN, Dedrick GS, Sizer PS, James CR. Changes in spinal height following sustained lumbar flexion and extension postures: a clinical measure of intervertebral disc hydration using stadiometry. J Manipulative Physiol Ther. 2009;32:358-63.
- 38. Page P. Current Concepts in Muscle Stretching for Exercise and Rehabilitation. Int J Sports Phys Ther. 2012;7:109-119.
- 39. Pape JL, Brismee JM, Sizer PS. Increased spinal height using propped slouched sitting postures: Innovative ways to rehydrate intervertebral discs.

- Appl Ergon. 2018;66:9-17.
- 40. Peterson T, Christensen R, Juhl C. Predicting a clinically important outcome in patients with low back pain following McKenzie therapy or spinal manipulation: a stratified analysis in a randomized controlled trial. BMC Musculoskelet Disord. 2015;74:1-7.
- 41. Puntumetakul R, Trott P, Williams M, Fulton I. Effect of time of day on the vertical spinal creep response. Appl Ergon. 2009;40:33-8.
- 42. Rousseau MA, Bradford DS, Hadi TM, Pedersen KL, Lotz JC. The instant axis of rotation influences facet forces at L5/S1 during flexion/extension and lateral bending. Eur Spine J. 2006;15:299-307.
- 43. Sady P, Wortman M, Blanke D. Flexibility training: ballistic, static or proprioceptive neuromuscular facilitation? Arch Phys Med Rehabil. 1982;63:261-263.
- 44. Simmerman SM, Sizer PS, Dedrick GS, Apte GG, Brismee JM. Immediate changes in spinal height and pain after aquatic vertical traction in patients with persistent low back symptoms: a crossover clinical trial. PM R. 2011;3:447-457.
- 45. Stankovic R, Johnell O. Conservative treatment of acute low-back pain. A prospective randomized trial: McKenzie method of treatment versus patient education in "mini back school". Spine. 1990;15:120-123.
- 46. Stothart JP, McGill SM. Stadiometry: on measurement technique to reduce variability in spine shrinkage measurement. Clin Biomech. 2000;15:546-8.
- 47. Surkitt LD, Ford JJ, Hahne AJ, Pizzari T, McMeeken JM., Efficacy of directional preference management for low back pain: a systematic review. Phys Ther. 2012;92:652-665.
- 48. Swinkels A, Cochrane K, Burt A, Johnson L, Lunn T, Rees AS. Exercise interventions for non-specific low back pain: An overview of systematic reviews. Phys Ther Rev. 2009;14:247-259.
- 49. Tonosu J, Matsudaira K, Oka H, Okazaki H, Oshio T, Hanaoka I et al. A population approach to analyze the effectiveness of a back extension exercise "One Stretch" in patients with low back pain: A replication study. J Orthop Sci. 2016; 21:414-418.
- 50. Tyrrell AR, Troup JD. Circadian variation in stature and the effects of spinal loading. Spine. 1985;10:161-164.
- 51.US Department of Labor Bureau of Labor Statistics: Standing or walking versus sitting on the job in 2016 (March 01, 2017); <a href="https://www.bls.gov/opub/ted/2017/standing-or-walking-versus-sitting-on-the-job-in-2016.htm">https://www.bls.gov/opub/ted/2017/standing-or-walking-versus-sitting-on-the-job-in-2016.htm</a>; Accessed 12/08/2017.

- 52. Vaisy M, Gizzi L, Petzke F, Consmuller T, Pfingsten M, Falla D. Measurement of Lumbar Spine Functional Movement in Low Back Pain. Clin J Pain. 2015;31:876-885.
- 53. Werneke MW, Hart DL, Cutrone G et al. Association Between Directional Preference and Centralization in Patients With Low Back Pain. J Orthop Sports Phys Ther. 2011;41:22-31.
- 54. Werneke MW, Hart DL, Resnik L, Stratford PW, Reyes A. Centralization: Prevalence and Effect on Treatment Outcomes Using a Standardized Operation Definition and Measurement Method. J Orthop Sports Phys Ther. 2008;38:116-125.
- 55. Yarznbowicz R, Tao M, Owens A, Wlodarski M, Dolutan J. Pain pattern classification and directional preference are associated with clinical outcomes for patients with low back pain. J Man Manip Ther. 2018;26:18-24.



Figure 1: Flow chart of test positions and testing sequence





# Second Visit





Measurement 4

▼

Trunk Ext Measure 2 Using Inclinometers

**Figure 2**: Starting position for trunk extensions.



**Figure 3:** Sustained trunk extension position and end position of repetitive trunk extensions.












Figure 6: Home instructions for Repetitive Trunk Extension

### **STANDING REPETITIVE EXTENSIONS**

-Start by standing with your feet shoulder width apart and place your hands on your hips. Lean back to arch your back then return to starting position. (Lean back as far as you can tolerate with each repetition)

Sets: 1

Repetitions: 10 (Performed in 45 seconds, rest 15 seconds)

-Perform sets in succession <u>Frequency</u>: 5 times per day





### **STANDING SUSTAINED EXTENSIONS**

-Start by standing with your feet shoulder width apart and place your hands on your hips. Lean back to arch your back, HOLD for time listed below, then return to starting position. (Lean back as far as you can tolerate with each repetition)

<u>Sets</u>: 1

Repetitions: 1 (hold extension 45 seconds,

rest 15 seconds)

-Perform sets in succession

Frequency: Five times per day

## Figure 8: Home instructions

Continue to use your medications, including medications aimed at decreasing your pain, as prescribed by your primary healthcare provider/physician. Please avoid changing them during the follow-up two-week period.

We will ask you to complete a sheet recording home exercise compliance when you come to the second treatment session in about two weeks.

Thank you.

#### APPENDIX A

# Volunteers Needed for a Research Study!

Title of the study:

"IMMEDIATE EFFECT OF STANDING TRUNK EXTENSION POSTURES ON SPINAL HEIGHT AND CLINICAL OUTCOME MEASURES IN LOW BACK PAIN: A RANDOMIZED CLINICAL TRIAL"

The purpose of this research is **to help Physical Therapists better treat patients with low back pain** by understanding the effects of motion on spine height.

Volunteers between the ages of 18-80 who currently have low back and/or leg pain are needed to participate in a Physical Therapy study conducted by the

Texas Tech University Health Sciences Center

Other **requirements for participation** in the study:

- Ability to stand for 5 minutes
- Ability to sit for a minimum of 10 minutes,
- Currently have low back pain that rate in the range of 2-9 on 10-point pain rating scale
- Subjects MUST NOT: be pregnant, have history of back surgery, spinal fractures, spinal fusion or spinal instability, current infection, inflammatory disease, cancer or be engaged in legal compensation claims for their back symptoms.

Participation is FREE. You will be asked to attend two, 1- hour sessions in 2-week period.



To compensate you for your time, you will receive free 1-month membership to Hill Country Memorial Wellness Center in Fredericksburg, Texas.

Contact Jeremy Harrison, PT, DPT, COMT (830)997-2001 jeremy.harrison@ttuhsc.edu

# APPENDIX B PRE-SCREENING QUESTIONNAIRE LUMBAR PAIN STUDY

### Please answer the following questions:

- 1. Are you interested to participate in a research project related to low back pain and spinal growth in which you will be asked to come twice to our clinic and be evaluated and treated twice for a 2-week period? You will be evaluated and treated free of charge for two sessions only.

  Yes / No
- 2. Are you between the ages of 18 and 80 years old?
  - a. Yes
  - b. No
- 3. Are you able to stand for 5 minutes?
  - a. Yes
  - b. No
- 4. Are you able to sit for 10 minutes?
  - a. Yes
  - b. No
- 5. Do you experience low back and/or leg pain of at least 2/10 and less or equal to 9/10?
  - a. Yes
  - b. No
- 6. Do you have any history of spinal surgery and/or fractures within the last 6 months?
  - a. Yes
  - b. No
- 7. Do you have a current history of acute systemic infection, active inflammatory disease, or malignancy?
  - a. Yes
  - b. No
- 8. Do you have any history of spinal fusion or diagnosed by a physician with spinal instability?
  - a. Yes
  - b. No

- 9. Are you currently engaged in legal/compensation claims for your back symptoms?
  - a. Yes
  - b. No
- 10. Is there a possibility that you could be pregnant?
  - a. Yes
  - b. No

Which, if any of the following positions, helps to relieve your back pain?

- a. Sitting
- b. Sitting with support in your back
- c. Standing
- d. Standing backward bending of your back
- e. Other:
- f. No position seems to feel better than the other

| FRONT OFFICE USE ONLY | | |
|------------------------------------------------|-----|----|
| Diagnosis of Lumbar Pain and/or Radiculopathy: | Yes | No |
| Patient referral for Physical Therapy: | Yes | No |

### If you are interested to participate, contact

Jeremy Harrison, PT, DPT - Investigator (830) 997-2001 jeremy.harrison@ttuhsc.edu

## Questionnaire Key

The purpose of this questionnaire is to take the burden off of participating physicians who are assisting with patient recruitment for this study. Simply add this questionnaire with your normal intake forms for all patients who are seeing the physician for low back pain and leg pain.

| Patient can be included in the study if: |
|---|
| Questions 1-5 |
| All answered "YES" |
| Questions 6-10 |
| All answered "NO" |
| Office Use Only section |
| <ul> <li>Qualified for study inclusion YES / NO</li> </ul> |
| Study Number: |
| Referral contact information: |
| Janaanse Hamisaas DT DDT COMT |
| Jeremy Harrison, PT, DPT, COMT |
| Texas Tech University HSC |
| 830-997-2001 |

# APPENDIX C

# **Intake Questionnaire:**

# To be filled out by the participant:

| Date: | _ Time:am pm |
|---|---|
| Last Name: | _ First Name <u>:</u> |
| Phone # :(day)(evening)_ | (cell) |
| E-mail address: | |
| Age: Gender: M / F. | |
| Do you currently have (within the past 24 or burning in any of the of following areas apply) | |
| Low back symptoms | Y/N |
| Buttock symptoms | Y/N |
| Thigh symptoms | Y/N |
| Lower leg symptoms (below the knee) | Y/N |
| Foot symptoms | Y/N |
| Toe symptoms | Y/N |
| How long ago did your current episode of pa<br>years | in start?daysmonths |
| Do you take pain medications? Yes / No | |
| If yes, i. Name the pain medications_ | |
| ii. How many hours ago did you | ı take your last pain medication? |

# <u>Do you currently have any of the following: (please circle yes for all that apply)</u>

| Height: | inches | Weight: | lbs |
|---|---|---|---|
| For Office us | se only | | |
| Yes/No | Non-English speaking | | |
| Yes/No | Pain level reported at 0/10 | at time of testing (no pai | n) |
| Yes/No | Pain level reported above 9 | 9/10 on Numerical Pain S | Scale. |
| Yes/No | Diagnosis of cauda equina | syndrome | |
| Yes/No | Any unhealed bone fractur | e | |
| Yes/No | Current vertebral infection | ı | |
| Yes/No | Vertebral fractures | | |
| Yes/No | Pain in shoulders or neck | | |
| Yes/No | History of spinal fusion/sur | gery | |
| Yes/No | Neurological disorders suc<br>injury, spinal tumors | ch as multiple sclerosis, s | spinal cord |
| Yes/No | Inability to stand upright fo | r a minimum of 5 minute | s |
| Yes/No | Inability to sit for a minimu | um of 5 consecutive mi | nutes |

# APPENDIX D

| Date: | 1. | <u>/20</u> | | Tin | ne: | an | n | _pm | S | Study | #: | | _ |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Please fil<br>the numb | | | | | | | _ | | e pair | ı in yo | our <i>B</i> | ACK c | ircling |
| What is th | | _ | | - | - | nave e | experi | ienced | d in th | e last | 2 day | s in yo | ur <b>back</b> |
| | | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | |
| What is th | | <del></del> | | - | - | nave ( | exper | ience | d in th | ie last | : 2 day | /s in yo | our <b>back</b> |
| | No | o Pain | | | | Мос | derate l | Pain | | | ι | Inbearab | le Pain |
| | | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | |
| What is th | | | | - | - | | | perier | nced ii | n the l | last 2 | days ir | ı your |
| | No | o Pain | | | | Мос | derate l | Pain | | | ι | Inbearab | le Pain |
| | | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | |
| What is th | ne amo | unt of | pain | you a | re exp | perier | ncing | in you | ır <b>bac</b> | k <u>rigl</u> | nt nov | <u>v</u> ? | |
| | No | o Pain | | | | Мос | derate l | Pain | | | ι | Inbearab | le Pain |
| | | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | |

### APPENDIX E

| Date: | 1. | /20 | Time: _ | am _ | pm | Study #: _ |
|-------|----|-----|---------|------|----|------------|
|-------|----|-----|---------|------|----|------------|

Please shade in the area of lower-back and /or legs where you have symptoms today.

(Symptoms include: Pain, tingling, numbness)

Por favor marke el area de su espalda baja o piernas donde tiene sintomas, el dia de hoy.

(Sintomas incluir: Dolar, hormigueo, o entumecimiento.)



Please circle the appropriate number below showing how bad your pain is now: Por favor marque abajo el numero que mostra que malo su dolor es ahora mismo.

No pain 0 1 2 3 4 5 6 7 8 9 10 Worst possible pain Sin dolor Dolorsisimo

# APPENDIX F

| Date: | /. / <b>20</b> | Time: | _ | am | pm | Study | /#: <u>_</u> |
|---|---|---|---|---|---|---|---|
| Me | odified Oswestry Low Back Pain Disa | bility Questionnairea | | | | | |
| TL | : | iiiiiii- | | | t. h | bask main bas at | Control |
| VO. | is questionnaire has been designed to<br>ur ability to manage in everyday life | . Please answer every | nic | uestion | by placing a r | nark in the one box | that |
| be | st describes your condition today. W | le realize you may fee | el t | hat two | of the stateme | ents may describe y | |
| co | ndition, but please mark only the b | ox that most closely | des | scribes | your current | condition. | |
| ъ. | 1. T. ( ) ( | | 724 | | | | |
| | in Intensity I can tolerate the pain I have without h | | | ing<br>I can si | t in any chair as | s long as I like. | |
| ·- | pain medication. | | | | | vorite chair as long as | I like. |
| | The pain is bad, but I can manage with | out having | | Pain pr | events me from | sitting for more than | 1 hour. |
| | to take pain medication. | | | | | sitting for more than | Ĺ |
| _ | Pain medication provides me with confrom pain. | | п | 1/2 hou | | sitting for more than | |
| | Pain medication provides me with mo | | _ | 10 min | | sitting for more than | |
| | from pain. | | | Pain pr | revents me from | sitting at all. | |
| | Pain medication provides me with littl | | 74- | | | | |
| | from pain. Pain medication has no effect on my p | | | nding | and as long as I | want without increas | sed nain |
| 13- | Tam medication has no effect on my p | | | | | want, but it increase | |
| | rsonal Care (e.g., Washing, Dressing) | | | my pai | n. | | |
| Ц | I can take care of myself normally wit increased pain. | nout causing | ш | | | standing for more th | an |
| | I can take care of myself normally, but | t it increases | | 1 hour. | | standing for more th | an |
| | my pain. | | _ | 1/2 hou | | standing for more in | |
| | It is painful to take care of myself, and | l I am slow | | | | standing for more th | an |
| п | and careful. I need help, but I am able to manage n | noet of my | П | 10 min | 777.7.7 | -t 1:t -11 | |
| | personal care. | lost of my | _ | Pain pi | events me from | standing at all. | |
| | I need help every day in most aspects | | Sle | eping | | | |
| | I do not get dressed, I wash with diffic | | | | | me from sleeping wel | |
| | stay in bed. | | | | | y using pain medicat | |
| Lit | fting | | ш | 6 hours | | ication, I sleep less th | ian |
| | I can lift heavy weights without increa | sed pain. | | | | ication, I sleep less th | nan |
| | I can lift heavy weights, but it causes i | ncreased pain. | | 4 hours | | , | |
| | Pain prevents me from lifting heavy w | | | | | ication, I sleep less th | ian |
| | the floor, but I can manage if the weig<br>conveniently positioned (e.g., on a tab | | п | 2 hours | events me from | sleening at all | |
| | Pain prevents me from lifting heavy w | | _ | r am pi | events me nom | siceping at an. | |
| | I can manage light to medium weights | if they are | Soc | ial Life | | | |
| П | conveniently positioned. | | | | | al and does not increa | se |
| | I can lift only very light weights. I cannot lift or carry anything at all. | | П | my pai | | al, but it increases my | lavel |
| | Tomas and or ourly any ming at any | | _ | of pain | | ii, but it ilicreases my | ievei |
| | alking | | | | | participating in more | e |
| | Pain does not prevent me from walking | | _ | | | g., sports, dancing). | |
| _ | Pain prevents me from walking more t $(1 \text{ mile} = 1.6 \text{ km}).$ | | | | | going out very often<br>social life to my hom | |
| | Pain prevents me from walking more t | | | | | al life because of my | |
| | Pain prevents me from walking more t | han 1/4 mile. | | | | | 200 |
| | I can walk only with crutches or a can<br>I am in bed most of the time and have | | | | | | |
| _ | the toilet. | | Plo | ase con | nlete avestions | aire on other side. | |
| | | | | | r.on questionin | and our owner blue. | |

| Traveling ☐ I can travel anywhere without increased pain. ☐ I can travel anywhere, but it increases my pain. ☐ My pain restricts my travel over 2 hours. ☐ My pain restricts my travel to short necessary journeys under 1/2 hour. ☐ My pain prevents all travel except for visits to the physician / therapist or hospital. | Employment / Homemaking My normal homemaking / job activities do not cause pain. My normal homemaking / job activities increase my pain, but I can still perform all that is required of me. I can perform most of my homemaking / job duties, but pain prevents me from performing more physically stressful activities (e.g., lifting, vacuuming). Pain prevents me from doing anything but light duties. Pain prevents me from doing even light duties. Pain prevents me from performing any job or homemaking chores. |
|---|---|
| FOR OFFICE USE ONLY Score: /50 x 100 =% points | |
| Scoring: For each section the total possible score is 5: if the statement is marked it = 5. If all ten sections are completed the Example: 16 (total scored) 50 (total possible score) x 100 = 32% If one section is missed or not applicable the score is calculated to a section is missed or n | ne score is calculated as follows: 6 6 7 8 7 8 8 8 8 8 8 8 8 8 8 |
| Name: | Date: |

Source: Fritz JM, Irrgang JJ. A comparison of a modified Oswestry Low Back Pain Disability Questionnaire and the Quebec Back Pain Disability Scale. *Physical Therapy*. 2001;81:776-788.

<sup>a</sup>Modified by Fritz & Irrgang with permission of The Chartered Society of Physiotherapy, from Fairbanks JCT, Couper J, Davies JB, et al. The Oswestry Low Back Pain Disability Questionnaire. *Physiotherapy*. 1980;66:271-273.

### APPENDIX G

| Date: | 1. | /20 | Time: _ | am | pm | Study #: |
|-------|----|-----|---------|----|----|----------|
|-------|----|-----|---------|----|----|----------|

### Fear-Avoidance Beliefs Questionnaire (FABQ) Waddell et al (1993) Pain, 52 (1993) 157 - 168

Here are some of the things which other patients have told us about their pain. For each statement please circle any number from 0 to 6 to say how much physical activities such as bending, lifting, walking or driving affect or would affect *your* back pain.

| | Completely | | | Unsure | | | Completely |
|---|---|---|---|---|---|---|---|
| | disagree | | | | | | agree |
| 1. My pain was caused by physical activity | 0 | 1 | 2 | 3 | 4 | 5 | 6 |
| 2. Physical activity makes my pain worse | 0 | 1 | 2 | 3 | 4 | 5 | 6 |
| 3. Physical activity might harm my back | 0 | 1 | 2 | 3 | 4 | 5 | 6 |
| 4. I should not do physical activities which (might) make my pain worse | 0 | 1 | 2 | 3 | 4 | 5 | 6 |
| 5. I cannot do physical activities which (might) make my pain worse | 0 | 1 | 2 | 3 | 4 | 5 | 6 |

The following statements are about how your normal work affects or would affect your back pain

Completely Unsure Completely

| | Completely | | | Unsure | | | Completely |
|---|---|---|---|---|---|---|---|
| | disagree | | | | | | agree |
| 6. My pain was caused by my work or by an accident at work | 0 | 1 | 2 | 3 | 4 | 5 | 6 |
| 7. My work aggravated my pain | 0 | 1 | 2 | 3 | 4 | 5 | 6 |
| 8. I have a claim for compensation for my pain | 0 | 1 | 2 | 3 | 4 | 5 | 6 |
| 9. My work is too heavy for me | 0 | 1 | 2 | 3 | 4 | 5 | 6 |
| 10. My work makes or would make my pain worse | 0 | 1 | 2 | 3 | 4 | 5 | 6 |
| 11. My work might harm my back | 0 | 1 | 2 | 3 | 4 | 5 | 6 |
| 12. I should not do my normal work with my present pain | 0 | 1 | 2 | 3 | 4 | 5 | 6 |
| 13. I cannot do my normal work with my present pain | 0 | 1 | 2 | 3 | 4 | 5 | 6 |
| 14. I cannot do my normal work till my pain is treated | 0 | 1 | 2 | 3 | 4 | 5 | 6 |
| 15. I do not think that I will be back to my normal work within 3 months. | 0 | 1 | 2 | 3 | 4 | 5 | 6 |
| 16. I do not think that I will ever be able to go back to that work | 0 | 1 | 2 | 3 | 4 | 5 | 6 |

### Scoring

Scale 1: fear-avoidance beliefs about work – items 6, 7, 9, 10, 11, 12, 15.

Scale 2: fear-avoidance beliefs about physical activity – items 2, 3, 4, 5.

Source: Gordon Waddell, Mary Newton, Iain Henderson, Douglas Somerville and Chris J. Main, A Fear-Avoidance Beliefs Questionnaire (FABQ) and the role of fear-avoidance beliefs in chronic low back pain and disability, *Pain*, 52 (1993) 157 – 168, 166.

# APPENDIX H

# Body diagram with template for centralization

| Date: | 1. | /20 | Time: | am | pm | Study #: |
|-------|----|-----|-------|----|----|----------|

### Numeric Overlay Template to the Patient's Body Diagrams



# APPENDIX I

| Date: /. | <u>/20</u> Tin | ne:am ¡ | pm Study #: | |
|---|---|---|---|---|
| Please complete the following form regarding compliance with your exercises: | | | | |
| Standing trunk extension exercises | | | | |
| | I did the exercise<br>25% of the time | | I did the exercise<br>75% of the time | |
| Were the exercises of backward bending | | | | |
| Very helpful | Helpful | Neutral | Not helpful | Not helpful at all |